CLINICAL TRIAL: NCT03077126
Title: Feasibility Study of Ultrasound Elastography Detecting Prostate Cancer: A Pilot Study
Brief Title: Feasibility Study of Ultrasound Elastography Detecting Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-17294
Record Dates: First submitted 2017-03-02; First posted 2017-03-10 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: elastography; ultrasound; prostate; cancer screening
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sodium phosphate; Enema; Ultrasonography; Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-surgery Ultrasound (Other): Aixplorer® ShearWave Elastography (SWE™) Ultrasound. Participants will undergo ultrasound prep with Fleet Enema and ultrasound procedure at their pre-op visit one to two weeks before their standard of care prostatectomy.
  Interventions: Other: Fleet Enema; Device: Aixplorer® ShearWave Elastography (SWE™); Diagnostic Test: Pre-surgery Ultrasound; Procedure: Prostatectomy

INTERVENTIONS:
Other: Fleet Enema — Since a probe will be introduced into the participant's rectal area, participants will be instructed to give themself one regular Fleet enema.
  Other Names: enema
Device: Aixplorer® ShearWave Elastography (SWE™) — Pre-surgery ultrasound: Aixplorer® ShearWave Elastography (SWE™) Ultrasound System (made by SuperSonic Imagine, Inc.). The device is used transrectally. This device (ultrasound system) has been cleared by the United States Food and Drug Administration (FDA) for the indication for use as described in this consent form.
  Other Names: ultrasound device; probe
Diagnostic Test: Pre-surgery Ultrasound — The ultrasound procedure referenced above will be performed at the participant's pre-op visit one to two weeks before their surgery.
  Other Names: Aixplorer® ShearWave Elastography (SWE™); ultrasound elastography
Procedure: Prostatectomy — Participants will undergo radical prostatectomy as currently performed at our Moffitt Cancer Center. This procedure is performed under general anesthesia in the operating room. This is considered standard of care.
  Other Names: prostate surgery

SUMMARY:
The main purpose of this study is to determine the accuracy and feasibility (possibility) of Aixplorer® ShearWave Elastography (SWE™) Ultrasound System (made by SuperSonic Imagine, Inc.) for detecting prostate cancer in men undergoing radical prostatectomy.

DETAILED DESCRIPTION:
The point estimate and its 95% confidence interval will be calculated using the exact binominal method. Identification of suspicious cancer tissue in a 12 prostate zone schema: Participants will undergo USE: Aixplorer® ShearWave Elastography (SWE™), (SuperSonic Imagine). Areas of the prostate with high suspicion for harboring cancer will be recorded in a 12 zone prostate schema. For study purposes the prostate will be divided into Zone 1(Left Lateral Base), Zone 2 (Left Base), Zone 3 (Right Base), Zone 4 (Right Lateral Base), Zone 5 (Left Lateral Mid), Zone 6 (Left Mid), Zone 7 (Right Mide), Zone 8 (Right Lateral Mid), Zone 9 (Left Lateral Apex), Zone 10 (Left Apex), Zone 11 (Right Apex), Zone 12 (Right Lateral Apex).

ELIGIBILITY:
Inclusion Criteria:

* Men with prostate cancer who elect surgery as the primary treatment of their cancer and to be performed at the Moffitt Cancer Center.
* Biopsy confirmed prostate cancer with at least ten biopsies performed for diagnosis.
* Location of cancer specified in the pathology report.
* Pathology reviewed by Moffitt pathologist

Exclusion Criteria:

* Less than ten biopsies obtained at time of diagnosis.
* Location of cancer not specified.
* Pathology not reviewed by Moffitt pathologist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04-11 (Actual); Primary Completion 2015-06-29 (Actual); Study Completion 2015-09-18 (Actual)

PRIMARY OUTCOMES:
Rate of Correlation Between Ultrasound Results and Pathology Results | 6 months
  Investigators will correlate the pathology findings from the radical prostatectomy specimen with the data recorded from USE.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Pow-Sang, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/